CLINICAL TRIAL: NCT05767567
Title: Evaluating the Efficacy of a Brief Online Intervention Among Current Heavy Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HR-22/23-34937
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-03

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Check Your Drinking (CYD) (Experimental): The CYD is a brief online intervention designed to provide personalized normative feedback aimed at motivating reductions in drinking
  Interventions: Behavioral: Brief Check Your Drinking (CYD)
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Brief Check Your Drinking (CYD) — The CYD is a brief online intervention designed to provide personalized normative feedback aimed at motivating reductions in drinking
  Arms: Brief Check Your Drinking (CYD)

SUMMARY:
Unhealthy alcohol consumption is common in the UK and causes tremendous harm to the individual, as well as harm to others. A significant gap in providing alcohol support is that most people with unhealthy alcohol consumption will never receive advice to cut down on their drinking. However, many are interested in self-directed interventions to help them evaluate their drinking and to motivate reductions in alcohol use. One such promising intervention uses online personalised normative feedback (PNF) which compares a person's drinking with others in the general population of the same age and sex. PNF interventions are thought to work because many people with unhealthy alcohol consumption overestimate how much others drink. Multiple trials have demonstrated that providing PNF to people with unhealthy consumption reduces their alcohol use . While several UK websites do provide feedback on assessment of risk (e.g., Down Your Drink introductory section, Alcohol Change UK), there appears to be no online intervention that provides PNF for unhealthy alcohol consumption.

The major objective of this pilot project is to conduct a two-arm, parallel group randomised controlled trial (RCT) in which 1,318 participants recruited from the Prolific website who have identified themselves as drinking 14 or more units per week are randomly assigned to one of two groups - a) those who are offered a PNF report, and b) those in a no intervention comparator group. Participants in the comparator group will not be provided any intervention materials but will instead be given a list of the different components of the PNF feedback and will be asked to think about how useful they would find each of them. Follow-up assessment will occur at 1 and 6 months post-randomisation. The project is described as a pilot because it is a preliminary evaluation of the PNF intervention in a UK context.

ELIGIBILITY:
Inclusion Criteria:

1) score 8 or more on the AUDIT (indicating current unhealthy alcohol use); and 2) endorsed the attention check questions correctly.

Exclusion Criteria:

Not meeting these inclusion criteria forms the exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 867 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Number of drinks consumed during a typical week | Three months

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Available from the PI upon reasonable request.